CLINICAL TRIAL: NCT01986816
Title: Lap Gastric Bypass and Its Impact on Wheightloss, QoL and Economic Cost
Brief Title: Return on Investment on Lap Gastric Bypass Regarding Quality of Life
Acronym: ROI-LGBP
Status: Withdrawn | Type: Observational
Why Stopped: Investigaotr no longer at LU.
Sponsor: Lund University (Other)
Collaborators: Landstinget i Kalmar Län (Other)
Responsible Party: Principal Investigator, Johan Berggren, MD, Lund University
Other Study IDs: ROI-LGBP
Record Dates: First submitted 2013-11-11; First posted 2013-11-19 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Obesity
Keywords: Obesity; Bariatric surgery; Laparoscopic gastric bypass; Quality of life; QALY
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate the cost of treatment and adverse efffects therof corresponds to quality of life improvements and expected wheightloss.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35
* age 18-60 years

Exclusion Criteria:

* Prior bariatric surgery
* Prior gastric surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Populutaion af morbid obese patients with BMI of 35 or more eligible for bariatric surgery
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Significant wheigtloss | 1 year

SECONDARY OUTCOMES:
Quality of life improvement | 3 months and 12 months post surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Kalmar County Hospital, Kalmar, Kalmar County, Sweden